CLINICAL TRIAL: NCT02007759
Title: Randomized Treatment of Neuromuscular Electrical Stimulation (NMES) for Dysphagia in Neonates
Brief Title: Neuromuscular Electrical Stimulation (NMES) for Dysphagia in Neonates
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty with recruiting patients; poor quality of EMG
Sponsor: Sanford Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SH NMES for Dysphagia
Record Dates: First submitted 2013-10-14; First posted 2013-12-11 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2016-09

CONDITIONS: Dysphagia
Keywords: Dysphagia; neuromuscular electrical stimulation; NMES; Neonates; Vitalstim
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VitalStim (Experimental): This group will be assigned to the active VitalStim unit.
  Interventions: Device: VitalStim
- Sham VitalStim (Sham Comparator): This group will be assigned to the sham VitalStim unit.
  Interventions: Device: Sham VitalStim

INTERVENTIONS:
Device: VitalStim — This group will receive active VitalStim treatment.
  Arms: VitalStim
Device: Sham VitalStim — This group will receive a sham VitalStim intervention.
  Arms: Sham VitalStim

SUMMARY:
The purpose of this study is to evaluate if the use of Neuromuscular Electrical Stimulation (NMES) will provide a more efficient method of treating neonates with dysfunctional oral feeding such as dysphagia. This study will attempt to determine if NMES applied to neonates at 36-42 weeks post-conception age (PCA) will decrease the need for nasogastric tubes (NG) and gastrostomy tubes (G-TUBE). Increase the rate at which these neonates complete full oral feeds, improve their swallowing skills, increase oral intake of calories, and gain weight.

ELIGIBILITY:
Inclusion Criteria:

* Male or female.
* Meet diagnostic criteria for dysphagia symptoms using the NOMAS and a VFSS.
* Infants with intraventricular hemorrhage (IVH) and hypoxic events can be included.
* Infants taking less than 5-10% of target volume by mouth between the ages of 36-42 weeks PCA.
* Multiple swallows to clear bolus following suck that includes a desaturation <80% and bradycardia <80 bpm.
* Apnea spells during feeds.
* Aspiration or penetration by VFSS

Exclusion Criteria:

* Known neurologic or neurodegenerative disorders.
* Chromosomal anomalies and syndromes.
* Cleft lip or palate.
* Birth defects.
* Unresolved cutaneous rash at the area of electrode placement.
* Medical condition that is a contraindication to NMES.

Ages: 36 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2013-11; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Reduction in G-tube rate insertions for the treatment grouped compared to the sham group. | Over the course of the treatment time frame to discharge, 2 weeks to 8 weeks
Increased percent of subjects towards achieving full oral feedings earlier in the subject's dysphagia treatment. | Over the course of the treatment time frame to discharge, 2 weeks to 8 weeks
Increase the amount of formula volume taken at feedings from beginning to end of study. | 2 weeks
Earlier NG tube removal for the treatment group compared to the control group. | Over the course of the treatment time frame to discharge, 2 weeks to 8 weeks

SECONDARY OUTCOMES:
Improve swallowing skills as measured by videofluoroscopic swallowing study (VFSS) and the video swallow assessment worksheet. | 2 weeks
Decrease spells with oral feeds over the course of the study. | 2 weeks
Allow for healthy weight gain via improved feedings. | 2 weeks
Increase the caloric intake orally. | 2 weeks
Decrease the oxygen requirement before and after study. | 2 weeks
Decrease inpatient length of stay. | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Akram Khan, MD, Principal Investigator — Sanford Health
Locations (1):
- Sanford USD Medical Center, Sioux Falls, South Dakota, United States